CLINICAL TRIAL: NCT04920435
Title: Prediction of the Response to Neoadjuvant Radiation Chemotherapy Through Texture Analysis Derived From Magnetic Resonance Imaging, Contrast Injection Computed Tomography and Positron Emission Tomography at 18-FDG in Locally Advanced Rectal Cancer
Brief Title: Prediction of the Response to Neoadjuvant Radiation Chemotherapy Through Texture Analysis Derived From Medical Imaging
Acronym: RECTOMICS
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: RECTOMICS (29BRC20.0027)
Record Dates: First submitted 2021-06-03; First posted 2021-06-09 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-11

CONDITIONS: Rectal Cancer
Keywords: locally advanced rectal cancer; radiomic
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- training population: patients from which we will develop the prediction model
- testing population: patients on whom we will test the prediction model

SUMMARY:
In patient with complete pathological response, surgery could be omitted without compromising progression-free or overall survival. A powerful prediction model is needed to guide management of this population.

Radiomics features provide complementary information about tumor heterogenity.

The aim of the investigators is to develop a model combining clinical and radiomic criteria able to predict complete pathological response.

ELIGIBILITY:
Inclusion Criteria:

* locally advanced rectal cancer
* patients who received concomitant radio-chemotherapy followed by surgery
* pre-therapeutic MRI and CT-scan dicom available

Exclusion Criteria:

* age under 18 yo
* lack of MRI or CT-scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with locally advanced rectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Prediction of the complete response (pCR) to neoadjuvant chemoradiotherapy | TO = Immediately after biopsy and extension evaluation.
  defined as the absence of tumor residue on the surgical specimen, ypT0N0

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Centre Hospitalier de Cornouaille, Quimper, Brittany Region
  - ICO, Nantes, Saint Herblain
  - CHRU de Brest (Morvan), Brest

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning one year and ending five years following the publication
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.